CLINICAL TRIAL: NCT04290221
Title: Comparing Effectiveness Two Intratissue Percutaneous Electrolysis (EPI) Interventions for Chronic Low Back Pain: Lumbar Nerve Root Stimulation vs Trigger Points Stimulation
Brief Title: Effectiveness Analysis of Ultrasound-guided Intratissue Percutaneous Electrolysis (EPI) in Patient With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, Adelaida María Castro-Sánchez, PhD, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UALBIO2019/037
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2023-09

CONDITIONS: Chronic Low-back Pain
Keywords: Intratissue Percutaneous Electrolysis; Trigger points; Lumbar nerve root; Randomized clinical trial; Electrical dry needling

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percutaneous electrolysis in the lumbar nerv (Experimental): This group will be treated with intratissue percutaneous electrolysis using a needle G32 with galvanic current as a cathodic flow electrode in the posterior nerve root of L3, L4 and L5, bilaterally (one times per week / 6 weeks). The intervention will be guided by ultrasound equipment medically certified (Directive 93/42 / EEC) device (EPI Advanced Medicine, Barcelona, Spain).
  Interventions: Other: Ultrasound-guided percutaneous electrolysis in the lumbar nerve root
- Electrical dry needling in trigger points (Active Comparator): It consists in apply the electrical dry needling on active and/or latent TPs in the gluteus medius, quadratus lumborum, and erector spinae muscles of the subjects L3 (one times per week / 6 weeks).
  Interventions: Other: Electrical Dry Needling in trigger points

INTERVENTIONS:
Other: Ultrasound-guided percutaneous electrolysis in the lumbar nerve root — This group will be treated with intratissue percutaneous electrolysis using a needle G32 with galvanic current as a cathodic flow electrode in the posterior nerve root of L3 (one times per week / 6 weeks). The intervention will be guided by ultrasound equipment medically certified (Directive 93/42 / EEC) device (EPI Advanced Medicine, Barcelona, Spain).
  Arms: Percutaneous electrolysis in the lumbar nerv
Other: Electrical Dry Needling in trigger points — It consists in apply the ultrasound-guided percutaneous electrolysis on active and/or latent TPs in the gluteus medius, quadratus lumborum, and erector spinae muscles of the subjects L3 (one times per week / 6 weeks).
  Arms: Electrical dry needling in trigger points

SUMMARY:
The main objective of this study is to analyze the effectiveness of the lumbar nerve root stimulation with ultrasound-guided percutaneous electrolysis versus the electrical dry needling of trigger points in patients with chronic low back pain.

DETAILED DESCRIPTION:
Given that recently the effectiveness of intratissue percutaneous electrolysis (EPI) has become of interest in the treatment of chronic musculoskeletal pain, when conventional physiotherapy management is not successful, the EPI can promote the healing biological processes. Several studies have demonstrated that inflammation can play an important role in the progression of muscle degeneration, in addition to potentially contributing to painful symptoms in individuals with chronic low back pain.

This technique involves nonthermal, electrochemical ablation of the lesion via the use of a cathodic fluid. The inflammation provoked is very localized and healing is rapid. Although EPI has been widely employed lately, the literature contains few studies validating its use.

The good results reported in studies of tendinopathies have to the undertaking of the present work, which compares the long-term effectiveness of EPI and dry needling-both ultrasound-guided-for the treatment of chronic low back pain.

A double blind clinical trial will be developed in a sample of 80 subjects with chronic low back pain. Patients of experimental group will receive 1 weekly sessions of intratissue percutaneous electrolysis for 3 weeks, for a total of 3 sessions. The aim is to compare the effectiveness of applying percutaneous electrolysis in the lumbar nerve root versus applying electrical dry needling on trigger points of the gluteus medius, quadratus lumborum, and erector spinae muscles (6 sessions, once a week) on disability, pain, fear of movement, quality of life, resistance of the trunk flexors, lumbar mobility and muscular electrical activity.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain ≥ 3 months.
* Age between 30 and 67 years old.
* Score ≥ 4 points on the Roland Morris Disability Questionnaire.
* Not being receiving other physical therapy.

Exclusion Criteria:

* Presence of lumbar stenosis.
* Diagnosis of spondylolisthesis.
* Diagnosis of fibromyalgia.
* Treatment with corticosteroids or oral medication in recent weeks.
* History of spine surgery.
* Contraindication of analgesic electrical therapy.
* Have previously received a treatment of intratissue percutaneous electrolysis.
* Central or peripheral nervous system disease.

Ages: 30 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2023-06-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Algometry | At baseline, at 3 weeks, at 6 weeks, and 1 month after the last intervention.
  An instrument for measuring the degree of sensitivity to pain. We will carry out a location of the myofascial trigger points following the illustrations of location of the myofascial trigger points that indicate Travell and Simons of both the left and right hemibody.
  Once located they will be classified as active or latent. Measured in kg / cm 2 with an analog pressure algometer model Wagner FDK20. To carry out this diagnosis using the analog pressure algometer, a force of 1Kg / sec will be applied until the subject indicates with a "YA" presence of pain, at that time we will stop the pressure made with the analog pressure algometer and record the result. The measurement will be executed 3 times with a 30 sec rest between each measurement and an average of the 3 results obtained will be obtained.
  Myofascial trigger points that do not meet the above criteria will be considered latent and which will not be subject to any treatment.
Change from baseline in Roland Morris Disability Questionnaire (RMDQ). | At baseline, at 3 weeks, at 6 weeks, and 1 month after the last intervention.
  This is a self-reported questionnaire consisting in 24 items reflecting limitations in different activities of daily living attributed to low back pain including walking, vending over, sitting, lying down, dressing, sleeping, self-care and daily activities.

SECONDARY OUTCOMES:
Change from baseline in disability. Oswestry Low Back Pain Disability Idex. | At baseline, at 3 weeks, at 6 weeks, and 1 month after the last intervention.
  It has 10 items associated to activities of daily living, each item has a punctuation from 0 to 5 points.
Change from baseline in pain intensity. Visual analogue scale. | At baseline, at 3 weeks, at 6 weeks, and 1 month after the last intervention.
  A 10-point Numerical Pain Scale (0: no pain, 10: maximum pain) assesses the intensity of pain
Change from baseline in Fear of Movement. Tampa Scale of kinesiophobia. | At baseline, at 3 weeks, at 6 weeks, and 1 month after the last intervention.
  Is a 17-item questionnaire that measures the fear of movement and (re)injury.
Change from baseline on Quality of Life. SF-36 Health questionnaire. | At baseline, at 3 weeks, at 6 weeks, and 1 month after the last intervention.
  SF-36 Health questionnaire scores range from 0 to 100% and indicate the self-perceived health-related quality of life.
Change from Mcquade Test. | At baseline, at 3 weeks, at 6 weeks, and 1 month after the last intervention.
  It measures the isometric endurance of trunk flexion muscles.
Change from baseline in range of motion and lumbar segmental mobility | At baseline, at 3 weeks, at 6 weeks, and 1 month after the last intervention.
  This variable is quantified using the SpinalMouse ® device (Phisiotech, Spain). It is an electronic computer-aided measuring device that measures sagittal spinal amplitude of movement (ROM) and intersegmental angles in a non-invasive way.
Change from baseline in Fingers-floor distance (cm) | At baseline, at 3 weeks, at 6 weeks, and 1 month after the last intervention.
  The patient flexes the trunk forward from the standing position, and the distance from the fingers to the ground is measured.
Change from baseline in Quality of Sleep . Pittsburgh Quality of Sleep Questionnaire Index | At baseline, at 3 weeks, at 6 weeks, and 1 month after the last intervention.
  The Pittsburgh Quality of Sleep Questionnaire Index (PSQI) will be used to study the quality of sleep. It comprises 24 items where the subjects respond to 19 of these items, and individual living in the same dwelling (or hospital room) responds to the remaining 5. Scores are obtained on each of 7 components of sleep quality: subjective quality, sleep latency, sleep duration, habitual sleep efficacy, sleep perturbations, use of hypnotic medication, and daily dysfunction.
Change from baseline in Anxiety. Hospital Anxiety and Depression Scale (HADS) | At baseline, at 3 weeks, at 6 weeks, and 1 month after the last intervention.
  The HADS is a 14-question instrument that measures anxiety and depression. Each question is scored between 0 (no impairment) and 3 (severe impairment), with a maximum score of 21 for anxiety or depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Almeria, Almería, Almeria, Spain

REFERENCES:
- [Background] de Miguel Valtierra L, Salom Moreno J, Fernandez-de-Las-Penas C, Cleland JA, Arias-Buria JL. Ultrasound-Guided Application of Percutaneous Electrolysis as an Adjunct to Exercise and Manual Therapy for Subacromial Pain Syndrome: A Randomized Clinical Trial. J Pain. 2018 Oct;19(10):1201-1210. doi: 10.1016/j.jpain.2018.04.017. Epub 2018 May 16. PMID 29777953
- [Background] Freeman MD, Woodham MA, Woodham AW. The role of the lumbar multifidus in chronic low back pain: a review. PM R. 2010 Feb;2(2):142-6; quiz 1 p following 167. doi: 10.1016/j.pmrj.2009.11.006. PMID 20193941
- [Background] Shahidi B, Hubbard JC, Gibbons MC, Ruoss S, Zlomislic V, Allen RT, Garfin SR, Ward SR. Lumbar multifidus muscle degenerates in individuals with chronic degenerative lumbar spine pathology. J Orthop Res. 2017 Dec;35(12):2700-2706. doi: 10.1002/jor.23597. Epub 2017 May 23. PMID 28480978
- [Background] Shahidi B, Parra CL, Berry DB, Hubbard JC, Gombatto S, Zlomislic V, Allen RT, Hughes-Austin J, Garfin S, Ward SR. Contribution of Lumbar Spine Pathology and Age to Paraspinal Muscle Size and Fatty Infiltration. Spine (Phila Pa 1976). 2017 Apr 15;42(8):616-623. doi: 10.1097/BRS.0000000000001848. PMID 27517512
- [Background] Abat F, Gelber PE, Polidori F, Monllau JC, Sanchez-Ibanez JM. Clinical results after ultrasound-guided intratissue percutaneous electrolysis (EPI(R)) and eccentric exercise in the treatment of patellar tendinopathy. Knee Surg Sports Traumatol Arthrosc. 2015 Apr;23(4):1046-52. doi: 10.1007/s00167-014-2855-2. Epub 2014 Jan 30. PMID 24477495
- [Background] Tuzun EH, Gildir S, Angin E, Tecer BH, Dana KO, Malkoc M. Effectiveness of dry needling versus a classical physiotherapy program in patients with chronic low-back pain: a single-blind, randomized, controlled trial. J Phys Ther Sci. 2017 Sep;29(9):1502-1509. doi: 10.1589/jpts.29.1502. Epub 2017 Sep 15. PMID 28931976
- [Background] Iborra-Marcos A, Ramos-Alvarez JJ, Rodriguez-Fabian G, Del Castillo-Gonzalez F, Lopez-Roman A, Polo-Portes C, Villanueva-Martinez M. Intratissue Percutaneous Electrolysis vs Corticosteroid Infiltration for the Treatment of Plantar Fasciosis. Foot Ankle Int. 2018 Jun;39(6):704-711. doi: 10.1177/1071100718754421. Epub 2018 Feb 13. PMID 29436233
- [Background] Jensen TS, Karppinen J, Sorensen JS, Niinimaki J, Leboeuf-Yde C. Vertebral endplate signal changes (Modic change): a systematic literature review of prevalence and association with non-specific low back pain. Eur Spine J. 2008 Nov;17(11):1407-22. doi: 10.1007/s00586-008-0770-2. Epub 2008 Sep 12. PMID 18787845
- [Background] Shahidi B, Fisch KM, Gibbons MC, Ward SR. Increased Fibrogenic Gene Expression in Multifidus Muscles of Patients With Chronic Versus Acute Lumbar Spine Pathology. Spine (Phila Pa 1976). 2020 Feb 15;45(4):E189-E195. doi: 10.1097/BRS.0000000000003243. PMID 31513095
- [Background] Goubert D, Oosterwijck JV, Meeus M, Danneels L. Structural Changes of Lumbar Muscles in Non-specific Low Back Pain: A Systematic Review. Pain Physician. 2016 Sep-Oct;19(7):E985-E1000. PMID 27676689
- [Background] Arias-Buria JL, Truyols-Dominguez S, Valero-Alcaide R, Salom-Moreno J, Atin-Arratibel MA, Fernandez-de-Las-Penas C. Ultrasound-Guided Percutaneous Electrolysis and Eccentric Exercises for Subacromial Pain Syndrome: A Randomized Clinical Trial. Evid Based Complement Alternat Med. 2015;2015:315219. doi: 10.1155/2015/315219. Epub 2015 Nov 15. PMID 26649058
- [Background] Valera-Garrido F, Minaya-Munoz F, Medina-Mirapeix F. Ultrasound-guided percutaneous needle electrolysis in chronic lateral epicondylitis: short-term and long-term results. Acupunct Med. 2014 Dec;32(6):446-54. doi: 10.1136/acupmed-2014-010619. Epub 2014 Aug 13. PMID 25122629